CLINICAL TRIAL: NCT03127657
Title: Effect of Cock's Comb Extract in the Treatment of Arsenical Skin Lesion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU-011-CT
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Chronic Arsenic Poisoning

STUDY DESIGN:
Intervention Model Description: Topical application of cock's comb extract in the treatment of palmar arsenical keratosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cock's comb extract 0.01% (Experimental): 25 Patients Cock's comb extract 0.01% Applied topically twice daily for 12 weeks
  Interventions: Drug: Cock's comb extract 0.01%

INTERVENTIONS:
Drug: Cock's comb extract 0.01% — Applied topically twice daily for 12 weeks
  Other Names: Cock's comb extract cream

SUMMARY:
Cock's comb extract is rich in hyaluronic acid, which is used as viscosupplementation injection and oral supplementation for osteoarthritis. Hyaluronic acid acts as humectants and topical moisturizing agent to the skin due to excellent moisturizing property. It has anti-inflammatory effect and used in the treatment of ulcer healing and to reduce the intensity of radioepithelitis. It is also used as a topical vehicle for the delivery of drug to the skin in actinic keratosis. In the case of arsenical keratotic nodule, topical application of hyaluronic acid may tends to decrease keratosis by repeated hydration of the skin. Therefore, the study will be conducted to determine any beneficial effect of topical application of cock's comb extract in the treatment of the patients with severe palmar arsenical keratosis.

DETAILED DESCRIPTION:
Cock's comb extract is rich in hyaluronic acid, which is used as viscosupplementation injection and oral supplementation for osteoarthritis. Hyaluronic acid is extensively utilized in many cosmetic products because of its moisturizing property as a topical moisturizing agent. It is also used as dermal fillers for wrinkle correction. It has anti-inflammatory effect and used in the treatment of different type of ulcers. In case of acute radioepithelitis, 0.2% hyaluronic acid is used to reduce inflammation. Hyaluronic acid has found important application in drug delivery system. Recently 3% diclofenac in 2.5% hyaluronic acid gel has been approved for the treatment of actinic keratoses as a unique topical vehicle for the localized delivery of drug to the skin. It is also used as a vehicle for various anticancer drugs. As it has many effective topical applications, it can be used in arsenical keratosis. In the case of arsenical keratotic nodule, topical application of hyaluronic acid may cause repeated hydration of the skin as a result keratosis tends to soften and disappear. Therefore, the study will be conducted to identify the outcome of cock's comb extract in the treatment of arsenical skin lesion. Biological activity and cytotoxicity of cock's comb extract have been identified after performing brine shrimp bioassay test. Twenty-five patients with severe palmar (>5 mm) arsenical keratosis will be recruited on the basis of inclusion and exclusion criteria. Before the study, water and nail samples will be collected to confirm arsenicosis. Blood samples will be collected for liver and kidney function test to observe any adverse effects of topically applied cock's comb extract both before and after the study. The cream will be prepared with 0.01% cock's comb extract mixed with olive oil, bee wax and benzoic acid for topical application 2 days prior visit of the recruited patients. The patient will be applied the cream on the affected area with a clean fingertip by rubbing gently at twice daily for 12 weeks without any interruption. Primary parameters will be the measurement of keratotic nodular size by slide calipers and perception scoring of the patients by Likert scale before and 12 weeks after the study. Secondary parameters will be the measurement of arsenic level in drinking water and nails of the recruited patients.

ELIGIBILITY:
Inclusion Criteria: (Patients)

* Age: 18-60 years
* Sex: Both male and female
* Arsenical keratosis: Presence of severe keratosis (>5mm) in both palms
* Drinking arsenic contaminated water (>50 µg/L) for at least more than 6 months
* Patient voluntarily agreed to participate
* Patient who understood the instruction of applying drug and could apply drug as per as instruction

Exclusion Criteria:

* Age <18 and >60 years
* Pregnant and nursing mother
* Palmar psoriasis
* Eczema
* Any kind of systemic disease, inflammatory disease and infectious condition that affect skin for example diabetes mellitus, rheumatoid arthritis, systemic lupus erythrematosus, hepatitis
* Hypersensitivity to avain protein
* Malignancy
* Impaired renal function - if creatinine level >1.3 mg/dl incase of men and >1.1 mg/dl in case of women
* Patient who received any treatment of arsenicosis within last three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-01-17 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in palmer arsenical keratosis | [0 week (baseline), 12 weeks (end)] [ Safety Issue: No]] [Safety Issue: No]
  Size of keratotic lesion will be decreased

SECONDARY OUTCOMES:
Changes in arsenic level in nail | [0 week (baseline), 12 weeks (end)] [ Safety Issue: No]] [Safety Issue: Yes]
  Arsenic level in nail will be decreased

CONTACTS AND LOCATIONS:
Overall Officials: Fatema Chowdhury, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Shahrashti, Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No